CLINICAL TRIAL: NCT03287336
Title: Prevention of Postpartum Hemorrhage: Identifying Pregnant Women at Risk and Determining the Safe and Effective Use of Tranexamic Acid Using State-of-the-art Pharmacokinetic/Pharmacodynamics Modeling
Brief Title: Prevention of Postpartum Hemorrhage With Tranexamic Acid
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: George Washington University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH); National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, Homa K. Ahmadzia, PI, George Washington University
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Prevention
Other Study IDs: IND134701; UL1TR001876 (NIH); KL2TR001877 (NIH); K23HL141640 (NIH)
Record Dates: First submitted 2017-06-27; First posted 2017-09-19 (Actual); Results first posted 2025-03-25 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Postpartum Hemorrhage
Keywords: tranexamic acid; postpartum hemorrhage
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — Tranexamic Acid

STUDY DESIGN:
Intervention Model Description: Three doses of Tranexamic acid (5 mg/kg, 10 mg/kg, and 15 mg/kg) will be used in a dose escalation fashion by cohort with the lowest dose first.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (Experimental): Dose of Tranexamic acid 5mg/kg will be administered.
  Interventions: Drug: Tranexamic Acid
- Cohort 2 (Experimental): Dose of Tranexamic acid 10 mg/kg will be administered.
  Interventions: Drug: Tranexamic Acid
- Cohort 3 (Experimental): Dose of Tranexamic acid 15 mg/kg will be administered.
  Interventions: Drug: Tranexamic Acid

INTERVENTIONS:
Drug: Tranexamic Acid — Tranexamic acid dosage (5 mg/kg, 10 mg/kg and 15 mg/kg) administered in a dose escalating fashion by cohort with the lowest dose first.
  Other Names: TXA; Cyklokapron

SUMMARY:
Postpartum hemorrhage is a significant contributor to maternal morbidity and mortality and is worldwide. TXA has recently been proven to reduce mortality when given to women in setting of diagnosed PPH. US obstetricians and anesthesiologists are hesitant to use TXA in the peripartum period especially for prevention of PPH due to uncertainty of an optimal dose and safety profile. The purpose of this study is to characterize the pharmacokinetics of TXA when given prophylactically at time of delivery. In addition investigators will determine the pharmacodynamics of TXA in the peripartum period.

DETAILED DESCRIPTION:
Conduct a prospective, open-label, dose finding PK study in 30 pregnant 3rd trimester women scheduled for non-emergent cesarean section who are at risk for hemorrhage. Three doses of the drug will be administered in an escalating fashion by cohort with the lowest dose first. A maximum of 1 gram will be administered. TXA serum levels at several time points after delivery will be assayed. A PK model will be constructed for determining the optimal TXA dose administered at parturition.

ELIGIBILITY:
Inclusion Criteria:

* Women who are undergoing medically indicated cesarean section at greater than 34+0 weeks gestation or women undergoing elective cesarean section at 39+0 weeks gestation in accordance with recommendations from the American Congress of Obstetricians and Gynecologists
* Pregnant women with normal serum creatinine (serum creatinine < 0.9)
* Women between the ages of 18 and 50 years old

Exclusion Criteria:

* Patients younger than 18 or older than 50
* women with active thrombotic or thromboembolic disease
* Women with a history of arterial or venous thromboembolic event
* Women with inherited thrombophilia or preexisting conditions that predisposes them to thromboembolic events (i.e. lupus, antiphospholipid syndrome)
* Women with a subarachnoid hemorrhage
* Women with acquired defective color vision
* history of seizure disorder
* known renal dysfunction
* multiple gestations (Twin or triplet pregnancies)
* Hypersensitivity to Tranexamic acid or anti-fibrinolytic therapy
* History of liver dysfunction

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant women in 3rd trimester of pregnancy
Enrollment: 43 (Actual)
Dates: Start 2018-01-02 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Homa Ahmadzia, MD, Principal Investigator — George Washington University
Locations (1):
- James Slota, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ahmadzia HK, Luban NLC, Li S, Guo D, Miszta A, Gobburu JVS, Berger JS, James AH, Wolberg AS, van den Anker J. Optimal use of intravenous tranexamic acid for hemorrhage prevention in pregnant women. Am J Obstet Gynecol. 2021 Jul;225(1):85.e1-85.e11. doi: 10.1016/j.ajog.2020.11.035. Epub 2020 Nov 26. PMID 33248975

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Started | 13 | 15 | 15
Completed | 10 | 10 | 10
Not Completed | 3 | 5 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Total
Number analyzed (Participants) | 10 | 10 | 10 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 10 | 30
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] | 34 [25 to 40] | 31 [24 to 38] | 33 [23 to 41] | 33 [23 to 41]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 10 | 30
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 1
  Not Hispanic or Latino | 9 | 10 | 10 | 29
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 5 | 5 | 6 | 16
  White | 5 | 4 | 3 | 12
  More than one race | 0 | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 10 | 30

OUTCOME MEASURES:

1. Primary Outcome: PK Model Parameter Estimates
Description: Data obtained from assays of TXA in blood, dose group and patient characteristics; parameter estimates in 2 compartment model includes the clearance of the drug (L/hr).
Time Frame: Different time points ranging from surgery (T0) to 1 day postpartum.
Population: Groups are combined because in PKPD modeling the best model parameter estimates are determined from combination of individual participant data of the dose administered, patient characteristics, times of administration and drug level in plasma.
Measure: Geometric Mean (Standard Deviation); unit: L/hr
Groups:
- 5mg/kg: Dose group 1
- 10 mg/kg: Dose group 2
- 15 mg/kg: Dose group 3
Arm/Group | 5mg/kg | 10 mg/kg | 15 mg/kg
Number analyzed (Participants) | 10 | 10 | 10
L/hr | 8.85 (2.24) | 10.39 (2.62) | 9.45 (2.37)

2. Primary Outcome: Pharmacodynamics of Tranexamic Acid
Description: PD model parameters included concentration of TXA causing 50% of maximal fractional inhibition (IC50).
Time Frame: Different time points ranging from surgery (T0) to 1 day postpartum.
Population: Groups are combined because in PKPD modeling the best model parameter estimates are determined from combination of individual participant data of the dose administered, patient characteristics, times of administration and measured ML levels in plasma.
Measure: Geometric Mean (Standard Deviation); unit: mg/L
Groups:
- 5 mg/kg: Dose group 1
Arm/Group | 5 mg/kg | 10 mg/kg | 15 mg/kg
Number analyzed (Participants) | 10 | 10 | 10
mg/L | 5.49 (2.35) | 6.49 (2.88) | 9.45 (3.55)

3. Secondary Outcome: Estimated Blood Loss
Description: Intraoperative blood loss
Time Frame: During surgery
Measure: Median (Full Range); unit: mL
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 10 | 10 | 10
mL | 750 [600 to 2000] | 750 [518 to 1000] | 700 [400 to 800]

4. Secondary Outcome: Safety Parameters
Description: Safety parameters such as adverse events (including nausea/vomiting) and serious adverse events
Time Frame: During surgery, after surgery while in hospital, 2 weeks and 6 weeks postpartum
Measure: Number; unit: events
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 10 | 10 | 10
events | 9 | 8 | 6

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 9/10 | 8/10 | 6/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=10) | Cohort 2 (N=10) | Cohort 3 (N=10)
nausea and vomiting (Gastrointestinal disorders) | 8 | 6 | 4
itching (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
bradycardia (Cardiac disorders) | 0 | 1 | 0
blood in neonate's stool (Gastrointestinal disorders) | 0 | 0 | 1
neonatal thrombosis (Blood and lymphatic system disorders) | 0 | 0 | 1
facial rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2018-08-09): https://cdn.clinicaltrials.gov/large-docs/36/NCT03287336/Prot_004.pdf
  • Statistical Analysis Plan (2023-10-27): https://cdn.clinicaltrials.gov/large-docs/36/NCT03287336/SAP_005.pdf
  • Informed Consent Form (2019-02-06): https://cdn.clinicaltrials.gov/large-docs/36/NCT03287336/ICF_002.pdf